CLINICAL TRIAL: NCT03644745
Title: Integrated Web-Based Customer Engagement, Physical Exercise, and Coaching Platform for Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R43AG057337 (NIH)
Record Dates: First submitted 2017-08-15; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2017-08

CONDITIONS: Aging
Keywords: Aging

STUDY DESIGN:
Intervention Model Description: The first 5 volunteers will be assigned for the preliminary in-home deployment to test the usability and provide feedback to potentially refine the system. Researchers will provide each participant with an activity tracker and download the required software on the participant's computer and smart phone. After 1 week, two researchers will conduct a home visit to provide the participant with a brief introduction to the system. Participants will interact with the system for 30 days while researchers use protocol analysis to record usability issues. All interactions with the system will be recorded. After 30 days, we will conduct an interview with the participant designed to uncover issues. The outcome measures described below will also be recorded. After necessary changes to the engagement and coaching system are made, we will deploy the system in an additional 15 homes for 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VM @ Home Usability (Experimental): We will pilot our customer engagement and physical exercise system in the homes of up to 20 participants for 3 months. Participants will interact with the system on their own computers, smart phones, and/or televisions and wear an activity tracker throughout the study. Interactions include physical exercise, system usage, and video conferencing.
  Interventions: Behavioral: VM @ Home Usability

INTERVENTIONS:
Behavioral: VM @ Home Usability — Our primary outcome measures will be use of the coaching system features, level of daily physical activity, mood, self-efficacy, and user satisfaction. Secondary outcomes that will inform our further development and be important outcomes in subsequent trials include user adherence to their coaching goals, physical function and level of socialization. For the pilot study, we plan to assess physical function and level of socialization at baseline and at the end of 3 months. For the other outcome measures, we will be able to integrate the data collection into the VM@Home platform and coaching process.

SUMMARY:
The fast-growing older population coupled with the worsening shortage of caregivers and nurses will soon present our nation with severe societal and economic challenges. Older adults often struggle to maintain quality of life and independence in the presence of chronic diseases and isolation. Physical exercise and socialization have been shown to reduce chronic disease, depression, falls and to improve quality of life in older adults. Motivation and feedback are essential to continued engagement in a wellness program, but doing so through the traditional manner of in-person coaching can be prohibitively expensive. Vigorous Mind (VM) has been providing a web-based platform to promote sustained engagement in older adults primarily in senior living facilities. The platform provides dynamic and tailored content including reminiscence activities, favorite music and video, adaptive computer games and communication. With the help of the Consortium on Technology for Proactive Care, the investigators will enhance the current VM system with an additional interactive physical exercise module and a health coach with automated tailored messaging and incentives for continued engagement and adherence. This will optimize the VM system for home-based deployment, thus expanding the reach and impact of VM to potentially delay or even prevent institutionalization among older adults living independently.

DETAILED DESCRIPTION:
The goal of the proposed project is to test the feasibility of deploying an economically feasible, machine-assisted, home-based wellness coaching system for older adults. Our approach consists of four sub-phases: (1) development, (2) usability, (3) preliminary deployment, and (4) pilot evaluation and analysis. The investigators estimate that the investigators will complete this project plan within 9 calendar months.

Sub-phase 1: Development [3 months and 3 weeks]. During sub-phase 1, the investigators will focus on software development activities at both VM and NU. There are 2 deliverables resulting from this sub-phase:

Build coaching interface. VM has an administrator interface that facilitates the design, assignment to users and adherence monitoring of a cognitive exercise plan. Using NU's experience and expertise, our developers will broaden the VM functionality to include a physical exercise module that allows assignment of exercise plans to users, monitoring of users' adherence and social interactions, as well as the delivery of tailored feedback and encouragement. The reward system of VM which currently rewards engagement in a variety of activities will be adapted to also reward physical activity. VM will create a new user type for the coach that allows for data sharing and an ability to communicate with family and/or caregivers in addition to the participant.

Integrate GymCentral into VM. Developed by researchers at the University of Trento in Italy (an international member of the CTPC), the primary software developer is now a postdoctoral fellow at NU and key personnel on this grant application. GymCentral is a virtual training platform (virtual gym) specifically designed for older adults. The virtual gym delivers video exercises in a "classroom" where trainees can see the presence of other trainees as avatars and communicate with them. The virtual gym aims to boost older adults' social interaction and motivate them to adhere to physical exercises. Our team of developers will integrate this system with the VM platform so that GymCentral can be deployed and collect engagement data within the VM system.

Sub phase 2: Usability [1 month]. In sub-phase 2, VM will connect with several of its independent living community's clients that have agreed to help recruit 5 independently living older adults who have and use computers for a pilot study (recruiting details specified below). This group will serve as the early usability testers for the home version of the VM system (VM@Home) and provide iterative feedback for our developers. Each of these 5 individuals will be given VM@Home to use on their home computers for one month. During this month, each participant will be provided a wearable wrist accelerometer (e.g., Misfit), along with training on the devices and on VM@Home, engage regularly with the platform, and be contacted weekly by a health coach. The investigators plan to use an innovative remote usability testing approach developed and tested by our collaborator Dr. Jimison. The developer and tester team will periodically contact the participants, especially if any anomalies are detected. During the remote sessions, participants will be asked to interact with the VM modules (calendaring, messaging, brain games, and Web entertainment) and the new physical exercise module. The iterative usability feedback will be used to adapt the design of the system for deployment in Sub-phase 3.

Sub-phase 3: Pilot Test [3 months]. After usability testing has been completed and necessary changes implemented, the investigators will ramp up recruitment activities through existing VM clients who have agreed to participate in the study with the goal of deploying VM@Home in an additional 15 homes of independently living older adults in independent-living communities. The five individuals who were recruited for sub-phase 2 will be offered the opportunity to continue in the study as champions of the technology, for which the investigators will provide additional training and support. As champions, they will mentor those of the other 15 users who will need assistance. During this sub-phase, the investigators will measure system use (continuously), level of physical activity (daily from wearable), level of socialization (daily from monitoring and by survey at baseline and each month), and mood, self-efficacy, and user satisfaction all by self-report at baseline and each month.

At the end of the three months, the investigators will also debrief with each participant with a semi-structured interview to obtain overall feedback and suggestions. These debriefing sessions will help investigators and developers to enhance design specifications for a robust, reliable and effective integrated engagement and coaching system to provide guidance for the further development and testing in a much larger population in Phase II. This will include exploring best options for including reward systems for active participation.

Sub-phase 4: Analysis [1 month]. Although the investigators will be routinely analyzing the monitoring data from system use and daily activity feedback from the wearable activity tracker throughout the project for coaching purposes, the last month of the project will be devoted to analyzing the full set of primary and secondary outcomes, as well as the qualitative debriefing interviews. The results from this pilot will prepare us for a more expanded and more powerful intervention in our follow-on Phase II proposal.

ELIGIBILITY:
Inclusion Criteria:

* Living independently
* Able to read and speak English
* PCP approval to exercise
* Have a laptop PC or Windows based tablet
* Have WiFi in their home
* Have a smart phone with a data plan

Exclusion Criteria:

* Uncorrected vision or auditory impairment
* Cognitive impairment (MoCA<27)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in level of physical activity | At baseline (week 1) and again in the final week (week 12)
  Change in daily average number of steps from baseline week 1 to final week (up to 16 weeks, depending on trial phase) as measured by Fitbit

SECONDARY OUTCOMES:
Change in mood | At baseline (week 1) and again in the final week (week 12)
  Change in mood score from baseline to completion using PANAS
User satisfaction | Post participation (Week 12)
  User rated satisfaction with system as measured by the Client Satisfaction Questionnaire adapted to Internet-based interventions (CSQ-I)
Self-efficacy | At baseline (week 1) and again in the final week (week 12)
  Change in user rated self-efficacy as measured by the Generalized Self-Efficacy Scale
Adherence to goals | weekly (weeks 1-12)
  Change in percentage of cumulative assigned activity completion (number of minutes using/number of minutes scheduled) as measured by the VM@Home system
Level of socialization | At baseline (week 1) and again in the final week (week 12)
  Change in social network score, measured at baseline and again at the end of participation as measured by the Ludden Social Network Scale
Usability | Week 12
  Change in user rated usability and ease of use of system as measured by the Brooke System Usability Scale (1996)

CONTACTS AND LOCATIONS:
Overall Officials: Holly B Jimison, PhD, Study Director — Northeastern University; Yuval Malinsky, Principal Investigator — Vigorous Mind, Inc.
Locations (2):
- United States (2):
  - New Bridge on the Charles, Dedham, Massachusetts
  - Maplewood Senior Living, Weston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers. This is usability testing for a small business innovation award with a small study population; sharing data under these circumstances would be inappropriate.

REFERENCES:
- See also: Vigorous Mind, Inc. website — https://www.vigorousmind.com/
- See also: Consortium on Technology for Proactive Care (research group at Northeastern University) — http://ctpc.ccs.neu.edu/